CLINICAL TRIAL: NCT07302100
Title: Nutritional Status Assessment in Adult Patients Followed for Gastroenteropancreatic Neuroendocrine Tumors at Strasbourg University Hospital
Acronym: DENUTNE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9485
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor
Keywords: Gastroenteropancreatic Neuroendocrine Tumor; Neuroendocrine tumors; Gastroenteropancreatic; Gastrointestinal
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuroendocrine tumors represent a heterogeneous group of tumors, of which gastrointestinal (gastroenteropancreatic) NETs are the most frequent.

Therapeutic management involves several approaches: control of any secretory syndrome and tumor control. Surgery is the first-line treatment for localized stages. When there is distant metastasis, various systemic treatments can be combined or administered sequentially (somatostatin analogs, everolimus, sunitinib, radioablation, targeted internal radiotherapy, cytotoxic chemotherapy). Gastrointestinal NETs are most often well-differentiated and slow-growing tumors with a median overall survival of up to 9 years (all sites combined), making comprehensive management of these patients all the more important.

In the context of cancer management, malnutrition has been shown to be associated with a poorer prognosis. Similarly, addressing malnutrition and improving nutritional parameters have been associated with improved prognosis.

The impact of nutritional status in patients with slow-growing tumors such as gastrointestinal neuroendocrine tumors (NETs) is less well understood but could be a modifiable factor for improving quality of life and treatment efficacy.

The research hypothesis is that nutritional status is associated with the prognosis of patients with gastrointestinal NETs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years
* Patients being monitored for a digestive neuroendocrine tumor (gastric, pancreatic, intestinal), diagnosed between January 1, 2000, and November 30, 2024

Exclusion Criteria:

- Tumor reclassified as non-neuroendocrine by histopathology

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 to 70 years being monitored for a digestive neuroendocrine tumor (gastric, pancreatic, intestinal), diagnosed between January 1, 2000, and November 30, 2024
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Establish a proportion of patients with malnutrition | Up to 12 months
  The proportion of patients with malnutrition based on weight loss, compared to usual weight before the onset of illness, is distributed as follows:
  * weight loss ≥ 5% in 1 month or
  * weight loss ≥ 10% in 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Endocrinologie, Diabétologie, Nutrition - CHU de Strasbourg - France, Strasbourg, France